CLINICAL TRIAL: NCT06659848
Title: the Effect of Fasted Versus Post-meal HIIT on Glycemic Control in Men With Type 2 Diabetes Mellitus
Acronym: HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prince Sattam Bin Abdulaziz University (Other)
Responsible Party: Principal Investigator, Ahmad Saied Mohammad, Principal Investigator, Prince Sattam Bin Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCBR-352/2024; 2023/03/26426 (Other Grant/Funding Number: Prince Sattam Bin Abdulaziz University)
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Diabetes Mellitus; High Intensity Exercise; Glycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: A total of 160 men with T2DM were recruited from nearby hospitals and clinics to participate in this study and 123 completed the study follow-up. A licensed physician performed the preliminary evaluation for all participants. Participants were instructed to maintain their medications, their usual dietary habits and usual physical activity throughout the study period.
  Only men diagnosed with T2DM, aged 40-60 years and inactive (performing less than 150 min/week of moderate-intensity exercise for at least the last six months) were included in this study. Subjects treated with exogenous insulin, and those with cardiovascular or musculoskeletal diseases limiting participation in HIIT were excluded.
  Eligible subjects were randomly assigned to one of four groups. The Fasted-group practiced HIIT prebreakfast in the fasted state (8-12 h fasting). The Post-breakfast, Post-lunch and Post-dinner groups practiced HIIT 2h after breakfast, lunch, and dinner respectively. The primary outcome was gly
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Fasted-group (Experimental): practiced HIIT prebreakfast in the fasted state (8-12 h fasting)
  Interventions: Other: high intensity interval training
- Post-breakfast (Experimental): practiced HIIT 2 hours after breakfast
  Interventions: Other: high intensity interval training
- Post-lunch (Experimental): practiced HIIT 2 hours after lunch
  Interventions: Other: high intensity interval training
- Post-dinner (Experimental): practiced HIIT 2 hours after dinner
  Interventions: Other: high intensity interval training

INTERVENTIONS:
Other: high intensity interval training — The subjects in the four groups performed 12 weeks of supervised HIIE program on a motorized treadmill (h/p/cosmos, Pulsar 4.0, Nussdorf-Traunstein, Germany) with a rate of three sessions weekly. The session commenced with a 5 min warming-up and concluded with a 5 min cooling down period. The exercise effort component consisted of 5 intervals of HIIT. Each interval continues for four min of HIIT with exercise intensity ranging from 75% to 90% of the peak heart rate. Each active recovery period between exercise intervals included moderate exercise at intensity of 50% to 60% of the peak heart rate. Every 3 weeks, the exercise intensity was increased by 5% starting with 75% of the HRmax in the first 3 weeks, 80% in the following 3 weeks and progressed to 90% the HRmax in the last 3 weeks. The subject's heart rate throughout the HIIT session was monitored using a polar heart rate monitor (Polar, Kempele, Finland).

SUMMARY:
Background: Recently, high intensity interval training (HIIT) has emerged as a promising regimen for the management of type 2 diabetic subjects. However, there is no consensus on the best time for HIIT regarding nutritional status.

Purpose: to investigate the effect of fasted versus postprandial HIIT training on glycemic control in men with type 2 Diabetes Mellitus.

Methods: This study enrolled 123 subjects suffering from type 2 diabetes mellitus with ages between 40 and 60 years. Subjects were divided into 4 groups, The post-breakfast, post-lunch and post-dinner groups practiced HIIT 2h after breakfast, lunch, and dinner respectively. The HIIT program involved 3 sessions weekly for 12 weeks. Glycated hemoglobin, fasting blood glucose, fasting insulin, insulin sensitivity, body composition, and blood lipid values were evaluated pre- and post-intervention.

DETAILED DESCRIPTION:
METHODS Study Design This study was performed as a randomized, controlled trial and included four groups. The study procedures were carried out in the department of physical therapy and health rehabilitation, Prince Sattam Bin Abdulaziz University.

Ethical consideration The study protocol was approved by the Standing Committee of Bioethics Research in Prince Sattam bin Abdulaziz University, Saudi Arabia (ID: SCBR-352/2024). The study was conducted in line with the principles of the Declaration of Helsinki. All study participants have signed a written informed consent form. The aim, procedures and potential risks of the study were explained to the study population.

Participants:

A total of 160 men with T2DM were recruited from nearby hospitals and clinics to participate in this study and 123 completed the study follow-up. A licensed physician performed the preliminary evaluation for all participants. Participants were instructed to maintain their medications, their usual dietary habits and usual physical activity throughout the study period.

Only men diagnosed with T2DM, aged 40-60 years and inactive (performing less than 150 min/week of moderate-intensity exercise for at least the last six months) were included in this study. Subjects treated with exogenous insulin, and those with cardiovascular or musculoskeletal diseases limiting participation in HIIT were excluded.

Eligible subjects were randomly assigned to one of four groups. The Fasted-group practiced HIIT prebreakfast in the fasted state (8-12 h fasting). The Post-breakfast, Post-lunch and Post-dinner groups practiced HIIT 2h after breakfast, lunch, and dinner respectively. The primary outcome was glycated hemoglobin (HbA1c). Body composition, fasting blood glucose, fasting insulin, insulin resistance and lipid values were also evaluated. The experimental period was twelve weeks, and all outcomes were measured pre- and post-intervention period.

Sample size calculation The sample size was determined based on an estimated effect size (d = 0.40), derived from changes in HbA1c% observed in Al-Rawaf's study. To reject the null hypothesis, the probability was set at 0.05, with a power of analysis at 90%, calculated using G*power 3.0.10 software (University of Dusseldorf, Dusseldorf, Germany). A total of 96 participants were initially recruited. However, the sample size was increased to 125 to account for an anticipated dropout rate of up to 30%.

Anthropometrics assessments:

All participants were assessed for body weight and height. A weight and height scale (Detecto, made in USA) was used. Body mass index (BMI) was calculated using the following formula:

BMI = weight (kg) / height (m)2 The waist circumferences of all subjects were measured as per instruction. The body fat percentage of each subject was evaluated using InBody 770 multifrequency bioelectrical impedance analysis scale (BIA) (Biospace, Cerritos, California).

Blood sampling and analysis:

Pre- and post-intervention blood samples were obtained from all participants after 12hours overnight fast. Venous blood samples were collected from antecubital vein around 8:00 am. The collected samples were centrifuged at 4°C for 10 min and then stored at -80°C for further analysis. Blood samples were analyzed for glucose, lipid profile including total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, plasma triglycerides (Hitachi Automatic Analyzer 7600 Hitachi, Tokyo, Japan). HbA1c levels were measured using a Tosoh G7 automatic analyzer (Tosoh Bioscience, Tokyo, Japan). Serum insulin levels were measured by ECLIA using an E-Insulin kit (Roche Diagnostics, Mannheim, Germany). To exclude the potential acute effects of the last exercise bout, postintervention blood samples were collected 48-72 h after the last exercise session. Serum low-density lipoprotein (LDL) cholesterol levels were calculated using the Friedewald formula.

Exercise test In order to determine exercise training intensity all subjects underwent performed an incremental maximal cardiopulmonary exercise test according to standard Bruce protocol to determine the peak heart rate. A stationary CPET system (Quark CPET, COSMED, Italy) on a motorized treadmill (h/p/cosmos, Pulsar 4.0, Nussdorf-Traunstein, Germany) was used to perform the test. The flow sensor was calibrated using a 3.0-L syringe. CO2 and O2 sensors were calibrated against known gases before each test. The test was terminated when subjects reached the point of volitional exhaustion. Reaching peak effort was confirmed when respiratory gas exchange ratio was ≥1.10, in combination with dyspnea, and leg and/or general fatigue.

Exercise protocol The subjects in the four groups performed 12 weeks of supervised HIIE program on a motorized treadmill (h/p/cosmos, Pulsar 4.0, Nussdorf-Traunstein, Germany) with a rate of three sessions weekly. The session commenced with a 5 min warming-up and concluded with a 5 min cooling down period. The exercise effort component consisted of 5 intervals of HIIT. Each interval continues for four min of HIIT with exercise intensity ranging from 75% to 90% of the peak heart rate. Each active recovery period between exercise intervals included moderate exercise at intensity of 50% to 60% of the peak heart rate. Every 3 weeks, the exercise intensity was increased by 5% starting with 75% of the HRmax in the first 3 weeks, 80% in the following 3 weeks and progressed to 90% the HRmax in the last 3 weeks. The subject's heart rate throughout the HIIT session was monitored using a polar heart rate monitor (Polar, Kempele, Finland).

ELIGIBILITY:
Inclusion Criteria:

* Only men diagnosed with T2DM,
* Aged 40-60 years
* Inactive (performing less than 150 min/week of moderate-intensity exercise for at least the last six months)

Exclusion Criteria:

* Subjects treated with exogenous insulin
* Cardiovascular diseases limiting participation in HIIT
* Musculoskeletal diseases limiting participation in HIIT

Ages: 40 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2024-06-20 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-10-20 (Actual)

PRIMARY OUTCOMES:
Percentage of glycated hemoglobin | 3 months
  Percentage of glycated hemoglobin (HbA1c) levels are measured using a Tosoh G7 automatic analyzer (Tosoh Bioscience, Tokyo, Japan).

SECONDARY OUTCOMES:
Body weight in kg | 3 months
  All participants were assessed for body weight and height. A weight and height scale (Detecto, made in USA) was used.
Body Mass Index (BMI) in kg/m2 | 3 months
  Body mass index (BMI) was calculated using the following formula:
  BMI = weight (kg) / height (m)2
Waist Circumference in cm | 3 months
  The waist circumferences of all subjects were measured as per instruction.
Concentration of Fasting plasma insulin in μU/ml | 3 months
  Pre- and post-intervention blood samples were obtained from all participants after 12hours overnight fast. Venous blood samples were collected from antecubital vein around 8:00 am. The collected samples were centrifuged at 4°C for 10 min and then stored at -80°C for further analysis.
Concentration of Fasting blood glucose in mg/dl | 3 months
  Pre- and post-intervention blood samples were obtained from all participants after 12hours overnight fast. Venous blood samples were collected from antecubital vein around 8:00 am. The collected samples were centrifuged at 4°C for 10 min and then stored at -80°C for further analysis.
concentration of total blood cholesterol in mg/dl | 3 months
  Blood samples were analyzed for glucose, lipid profile including total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, plasma triglycerides (Hitachi Automatic Analyzer 7600 Hitachi, Tokyo, Japan).
concentration of total blood triglyceride in mg/dl | 3 months
  Blood samples were analyzed for glucose, lipid profile including total cholesterol, high-density lipoprotein (HDL) cholesterol, low-density lipoprotein (LDL) cholesterol, plasma triglycerides (Hitachi Automatic Analyzer 7600 Hitachi, Tokyo, Japan).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Ahmed, PhD, Principal Investigator — 1Department of Physical Therapy and Health Rehabilitation, College of Applied Medical Sciences, Prince Sattam bin Abdulaziz University, Al-Kharj, Saudi Arabia
Locations (1):
- Prince Sattam bin Abdulaziz University, Al Kharj, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
no need

REFERENCES:
- [Background] Mancilla R, Brouwers B, Schrauwen-Hinderling VB, Hesselink MKC, Hoeks J, Schrauwen P. Exercise training elicits superior metabolic effects when performed in the afternoon compared to morning in metabolically compromised humans. Physiol Rep. 2021 Jan;8(24):e14669. doi: 10.14814/phy2.14669. PMID 33356015
- [Background] Karstoft K, Winding K, Knudsen SH, Nielsen JS, Thomsen C, Pedersen BK, Solomon TP. The effects of free-living interval-walking training on glycemic control, body composition, and physical fitness in type 2 diabetic patients: a randomized, controlled trial. Diabetes Care. 2013 Feb;36(2):228-36. doi: 10.2337/dc12-0658. Epub 2012 Sep 21. PMID 23002086
- [Background] Madsen SM, Thorup AC, Overgaard K, Jeppesen PB. High Intensity Interval Training Improves Glycaemic Control and Pancreatic beta Cell Function of Type 2 Diabetes Patients. PLoS One. 2015 Aug 10;10(8):e0133286. doi: 10.1371/journal.pone.0133286. eCollection 2015. PMID 26258597
- [Background] Savikj M, Gabriel BM, Alm PS, Smith J, Caidahl K, Bjornholm M, Fritz T, Krook A, Zierath JR, Wallberg-Henriksson H. Afternoon exercise is more efficacious than morning exercise at improving blood glucose levels in individuals with type 2 diabetes: a randomised crossover trial. Diabetologia. 2019 Feb;62(2):233-237. doi: 10.1007/s00125-018-4767-z. Epub 2018 Nov 13. PMID 30426166
- [Background] Verboven K, Wens I, Vandenabeele F, Stevens AN, Celie B, Lapauw B, Dendale P, VAN Loon LJC, Calders P, Hansen D. Impact of Exercise-Nutritional State Interactions in Patients with Type 2 Diabetes. Med Sci Sports Exerc. 2020 Mar;52(3):720-728. doi: 10.1249/MSS.0000000000002165. PMID 31652237
- [Background] Nygaard H, Ronnestad BR, Hammarstrom D, Holmboe-Ottesen G, Hostmark AT. Effects of Exercise in the Fasted and Postprandial State on Interstitial Glucose in Hyperglycemic Individuals. J Sports Sci Med. 2017 Jun 1;16(2):254-263. eCollection 2017 Jun. PMID 28630579
- [Background] Peddie MC, Bone JL, Rehrer NJ, Skeaff CM, Gray AR, Perry TL. Breaking prolonged sitting reduces postprandial glycemia in healthy, normal-weight adults: a randomized crossover trial. Am J Clin Nutr. 2013 Aug;98(2):358-66. doi: 10.3945/ajcn.112.051763. Epub 2013 Jun 26. PMID 23803893
- [Background] Gillen JB, Little JP, Punthakee Z, Tarnopolsky MA, Riddell MC, Gibala MJ. Acute high-intensity interval exercise reduces the postprandial glucose response and prevalence of hyperglycaemia in patients with type 2 diabetes. Diabetes Obes Metab. 2012 Jun;14(6):575-7. doi: 10.1111/j.1463-1326.2012.01564.x. Epub 2012 Feb 20. PMID 22268455
- [Background] Hamasaki H. Daily physical activity and type 2 diabetes: A review. World J Diabetes. 2016 Jun 25;7(12):243-51. doi: 10.4239/wjd.v7.i12.243. PMID 27350847
- [Background] Kanaley JA, Colberg SR, Corcoran MH, Malin SK, Rodriguez NR, Crespo CJ, Kirwan JP, Zierath JR. Exercise/Physical Activity in Individuals with Type 2 Diabetes: A Consensus Statement from the American College of Sports Medicine. Med Sci Sports Exerc. 2022 Feb 1;54(2):353-368. doi: 10.1249/MSS.0000000000002800. PMID 35029593
- [Background] American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2021. Diabetes Care. 2021 Jan;44(Suppl 1):S15-S33. doi: 10.2337/dc21-S002. PMID 33298413
- [Background] Saeedi P, Petersohn I, Salpea P, Malanda B, Karuranga S, Unwin N, Colagiuri S, Guariguata L, Motala AA, Ogurtsova K, Shaw JE, Bright D, Williams R; IDF Diabetes Atlas Committee. Global and regional diabetes prevalence estimates for 2019 and projections for 2030 and 2045: Results from the International Diabetes Federation Diabetes Atlas, 9th edition. Diabetes Res Clin Pract. 2019 Nov;157:107843. doi: 10.1016/j.diabres.2019.107843. Epub 2019 Sep 10. PMID 31518657